CLINICAL TRIAL: NCT00354445
Title: A Phase IV, Open Label, Multi-Center, Study of Maintenance Intravitreous Injections of Macugen (Pegaptanib Sodium) Given Every 6 Weeks for 48 Weeks in Subjects With Subfoveal Neovascular Age-Related Macular Degeneration (AMD) Initially Treated With a Modality Resulting in Maculopathy Improvement
Brief Title: A Clinical Trial to Explore the Safety and Efficacy of Injections of Macugen When Given Every 6 Weeks in Subjects With AMD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eyetech Pharmaceuticals (Industry)
Collaborators: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EOP1023
Record Dates: First submitted 2006-07-18; First posted 2006-07-20 (Estimated); Last update posted 2007-01-15 (Estimated); Status verified 2007-01

CONDITIONS: Age-Related Macular Degeneration (AMD)
Keywords: Age-Related Macular Degeneration (AMD); pegaptanib sodium; subfoveal CNV; macugen
MeSH Terms: conditions — Macular Degeneration | interventions — pegaptanib

INTERVENTIONS:
Drug: pegaptanib sodium (Macugen)

SUMMARY:
The purpose of this study is to explore the safety and efficacy of Macugen given as maintenance therapy in patients who have had initial success with another AMD treatment. Patients must have 1, but not more than 3 prior treatments for Neovascular AMD.

ELIGIBILITY:
Inclusion Criteria:

* Subfoveal CNV secondary to AMD
* At least 1 but not more than 3 prior treatments for AMD

Exclusion Criteria:

* Subfoveal scar or subfoveal atrophy
* Significant media opacities, including cataract, which might interfere with visual acuity

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 2006-06

CONTACTS AND LOCATIONS:
Locations (1):
- Retina Research Institute of Texas, LLC, Abilene, Texas, United States

REFERENCES:
- [Derived] Friberg TR, Tolentino M; LEVEL Study Group; Weber P, Patel S, Campbell S, Goldbaum M. Pegaptanib sodium as maintenance therapy in neovascular age-related macular degeneration: the LEVEL study. Br J Ophthalmol. 2010 Dec;94(12):1611-7. doi: 10.1136/bjo.2009.174946. Epub 2010 May 14. PMID 20472746